CLINICAL TRIAL: NCT04594200
Title: Do Peer-comparisons, Emphasis on Harms, and/or Inclusion of Viral Prescription Pad Resources Increase Responsiveness to Feedback About Antibiotic Prescribing in Primary Care (PHO Trial)
Brief Title: Do Fair Comparisons or Harms Data Increase Responsiveness to Feedback About Antibiotic Prescribing: 2x2 Factorial Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Ontario Agency for Health Protection and Promotion (Other Government); College of Family Physicians of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Noah Ivers, Family Physician, Canada Research Chair (Tier 2) in Implementation of Evidence Based Practice, Women's College Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-0024-E (PHO Trial)
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Infection
Keywords: Antibiotics; Audit and Feedback
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: 2x2 Pragmatic Factorial Randomized Control Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intervention Group: Harms Emphasis - Simple Comparator (Experimental): Physicians in this group will receive a personalized antibiotic prescribing feedback letter which contains a simple comparator to represent a target or benchmark for antibiotic prescribing. For the simple comparator, we will rank the antibiotic prescribing outcomes for all Ontario family physicians and use the lowest quartile as the benchmark. The letter will also include information on both lack of benefit and potential harms caused by unnecessary use of antibiotics. Physicians will also receive a paper-copy viral prescription pad and will receive the intervention letter again 1-month post initial dissemination.
  Interventions: Behavioral: Audit and Feedback (A&F)
- Intervention Group: Harms Emphasis - Complex Comparator (Experimental): Physicians in this group will receive a personalized antibiotic prescribing feedback letter which contains a complex (adjusted) comparator to represent a target or benchmark for antibiotic prescribing. For the complex comparator, recipients will be compared only to top-performing 'like-peers' - the group of physicians with similar complexity and numbers of patients. We will adjust the prescribing indicators for patient sex, number of patients >85 years, rurality, continuity of care score, proportion of emergency room practice, proportion nursing home practice, neighborhood income quintile of patients, and rates of common patient comorbidities. The letter will also include information on both lack of benefit and potential harms caused by unnecessary use of antibiotics. Physicians will also receive a paper-copy viral prescription pad and will receive the intervention letter again 1-month later.
  Interventions: Behavioral: Audit and Feedback (A&F)
- Intervention Group: No Harms Emphasis - Simple Comparator (Experimental): Physicians in this group will receive a personalized antibiotic prescribing feedback letter which contains a simple comparator to represent a target or benchmark for antibiotic prescribing. For the simple comparator we will rank the antibiotic prescribing outcomes for all Ontario family physicians and use the lowest quartile as the benchmark. The letter will also include information on lack of benefit of unnecessary use of antibiotics. Physicians will also receive a paper-copy viral prescription pad and will receive the intervention letter again 1-month post initial dissemination.
  Interventions: Behavioral: Audit and Feedback (A&F)
- Intervention Group: No Harms Emphasis - Complex Comparator (Experimental): Physicians in this group will receive a personalized antibiotic prescribing feedback letter which contains a complex (adjusted) comparator to represent a target or benchmark for antibiotic prescribing. For the complex comparator, recipients will be compared only to top-performing 'like-peers' - the group of physicians with similar complexity and numbers of patients. We will adjust the prescribing indicators for patient sex, number of patients >85 years, rurality, continuity of care score, proportion of emergency room practice, proportion nursing home practice, neighborhood income quintile of patients, and rates of common patient comorbidities. The letter will also include information on lack of benefit of unnecessary use of antibiotics. Physicians will also receive a paper-copy viral prescription pad and will receive the intervention letter again 1-month later.
  Interventions: Behavioral: Audit and Feedback (A&F)
- Control Group (No Intervention): Participants in this group will not receive a personalized antibiotic prescribing feedback letter and they will not receive a viral prescription pad.

INTERVENTIONS:
Behavioral: Audit and Feedback (A&F) — In this protocol, we propose comparing 2 intervention design elements in a multifactorial design. Specifically, we will evaluate:
  i) an emphasis on antibiotic-associated harms in comparison to messages that focus on lack of benefit; ii) simple versus adjusted peer comparators to represent a target for the prescribing quality indicators
  We will also investigate the effects of the inclusion of materials developed by Choosing Wisely Canada (CWC) - namely the viral prescription pad - to help physicians act upon the feedback to reduce their prescribing
  Arms: Intervention Group: Harms Emphasis - Complex Comparator; Intervention Group: Harms Emphasis - Simple Comparator; Intervention Group: No Harms Emphasis - Complex Comparator; Intervention Group: No Harms Emphasis - Simple Comparator

SUMMARY:
Antibiotic overuse is common and antibiotic prescribing contributes to rising rates of antimicrobial resistance. Primary care physicians prescribe the majority of all antibiotics and there is large inter-physician variability in prescribing that cannot be explained by differences in patient populations.

Peer comparison audit and feedback (A&F) can act as an effective behavioural intervention to reduce unnecessary antibiotic use. The range of effects seen in prior A&F trials could be attributed, at least in part, to differences in the way the feedback interventions were designed. In fall 2018, the investigators conducted an audit and feedback trial of mailed letters to 3500 family physicians in Ontario who prescribe the highest volume of antibiotics [NCT03776383]. While effective, family physicians questioned the credibility of the report in terms of its ability to fairly account for their practice size and population.

In Ontario, A&F is routinely offered to primary care providers from a variety of sources. Ontario Health - an agency created by the Government of Ontario - provides A&F via email to physicians who voluntarily sign up for their "MyPractice" reports. These are multi-topic reports with aggregated (physician-level) data. As of November 2021, the MyPractice reports for family physicians will include data on antibiotic prescribing. To date, less than half of Ontario family physicians have signed up for the MyPractice reports from Ontario Health.

For this study, the investigators will conduct a trial to investigate the effect of A&F in family physicians not already receiving A&F through a MyPractice: Primary Care report. Physicians who do not already receive antibiotic prescribing feedback through a MyPractice report will receive personalized antibiotic prescribing feedback through a letter mailed out from PHO. This large-scale evaluation provides an opportunity to evaluate not only whether A&F using such data is helpful in the post-covid context, but how best to design the A&F intervention and to explore why we observed (or not) changes in antibiotic prescribing.

DETAILED DESCRIPTION:
This study will examine ways to optimize the effects of A&F for antibiotic prescribing in primary care. This study will aim to answer the following questions:

1. Do patients of family physicians receiving A&F about antibiotic prescribing receive fewer antibiotics compared to patients of family physicians that do not receive A&F?
2. Does the effects of A&F vary with the following design features? i) case-mix adjusted (or simple) peer comparators to represent a target for the prescribing quality indicators ii) emphasis (or not) on antibiotic-associated harms in addition to messages that focus on lack of benefit

This trial will include family physicians who did not opt-in to receive MyPractice: Primary Care report from Ontario Health. Physicians will be randomized to the control group or intervention group. Physicians in the intervention group will receive a personalized antibiotic prescribing feedback letter that will include personalized data regarding total antibiotic prescribing per 1000 patient visits and proportion of antibiotic prescriptions provided for a duration of >7 days. The letter will also contain two experimental factors: 1: Simple vs complex peer comparators; and 2) Emphasis or not on antibiotic harms. For the complex (adjusted) comparator, recipients will be compared only to top-performing 'like-peers' - the group of physicians with similar complexity and numbers of patients. For the harms vs no harms factor, physicians will be either provided with information that focuses on lack of benefit for certain conditions (no harms), or with information that emphasizes the potential harms caused by unnecessary use of antibiotics. The feedback letters will be mailed to each physicians' primary practice address, along with a viral prescription pad developed by Choosing Wisely Canada.

One month after the initial intervention, intervention participants will be invited to complete a process evaluation survey to determine why or why not the intervention worked and how individual factors can affect physician motivation, willingness, and ability to engage in new practices. Intervention participants will also be invited to take part in a process evaluation interview.

ELIGIBILITY:
Inclusion Criteria:

Family physicians with an active practice who prescribe antibiotics in Ontario to patients aged 65 or older.

Family physicians who did not sign up by September 2021 to receive the MyPractice report

Exclusion Criteria:

<100 unique patient visits in the most recent year or two of the three prior years for patients 65 years of age or older;

<10 antibiotic prescriptions to patients 65+ in the most recent year or two of the three prior years; or

previously opted out of antibiotic prescribing letters from PHO (n= 15)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5107 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescribing rate | 6 months
  total number of antibiotic prescriptions per 1000 65+ patient visits

SECONDARY OUTCOMES:
Proportion Antibiotic Rx with Prolonged Duration | 6 months
  antibiotics prescribed for more than 7 days per episode
Proportion Antibiotic Rx with Prolonged Duration | 12 months
  antibiotics prescribed for more than 7 days per episode
Antibiotic drug costs | 6 months
  Cost in CDN$
Antibiotic drug costs | 12 months
  Cost in CDN$
Antibiotics prescribed for viral infections | 6 months
  total number of antibiotic rx per 1000 65+ patient visits for presumed viral condition (and thus likely unnecessary) based on administrative database diagnostic codes
Antibiotics prescribed for viral infections | 12 months
  total number of antibiotic rx per 1000 65+ patient visits for presumed viral condition (and thus likely unnecessary) based on administrative database diagnostic codes
Total Antibiotic Days of Therapy | 6 months
  total number DOTs per 1000 65+ patient visits
Total Antibiotic Days of Therapy | 12 months
  total number DOTs per 1000 65+ patient visits
Proportion of broad spectrum antibiotic prescriptions | 6 months
  antibiotic prescriptions that are broad spectrum
Proportion of broad spectrum antibiotic prescriptions | 12 months
  antibiotic prescriptions that are broad spectrum

CONTACTS AND LOCATIONS:
Overall Officials: Noah M Ivers, Principal Investigator — WCH
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share this data.

REFERENCES:
- [Derived] Saqib K, Ivers N, Brown KA, Daneman N, Leung V, Langford BJ, Garber G, Grimshaw JM, Silverman MS, Taljaard M, Brehaut J, Thavorn K, Lacroix M, Friedman L, Shuldiner J, Gomes T, Gushue S, Leis JA, Zwarenstein M, Schwartz KL. Spillover From an Intervention on Antibiotic Prescribing for Family Physicians: A Post Hoc Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2518261. doi: 10.1001/jamanetworkopen.2025.18261. PMID 40591360
- [Derived] Shuldiner J, Lacroix M, Saragosa M, Reis C, Schwartz KL, Gushue S, Leung V, Grimshaw J, Silverman M, Thavorn K, Leis JA, Kidd M, Daneman N, Tradous M, Langford B, Morris AM, Lam J, Garber G, Brehaut J, Taljaard M, Greiver M, Ivers NM. Process evaluation of two large randomized controlled trials to understand factors influencing family physicians' use of antibiotic audit and feedback reports. Implement Sci. 2024 Sep 16;19(1):65. doi: 10.1186/s13012-024-01393-5. PMID 39285305
- [Derived] Schwartz KL, Shuldiner J, Langford BJ, Brown KA, Schultz SE, Leung V, Daneman N, Tadrous M, Witteman HO, Garber G, Grimshaw JM, Leis JA, Presseau J, Silverman MS, Taljaard M, Gomes T, Lacroix M, Brehaut J, Thavorn K, Gushue S, Friedman L, Zwarenstein M, Ivers N. Mailed feedback to primary care physicians on antibiotic prescribing for patients aged 65 years and older: pragmatic, factorial randomised controlled trial. BMJ. 2024 Jun 5;385:e079329. doi: 10.1136/bmj-2024-079329. PMID 38839101
- [Derived] Shuldiner J, Schwartz KL, Langford BJ, Ivers NM; Ontario Healthcare Implementation Laboratory study team. Optimizing responsiveness to feedback about antibiotic prescribing in primary care: protocol for two interrelated randomized implementation trials with embedded process evaluations. Implement Sci. 2022 Feb 14;17(1):17. doi: 10.1186/s13012-022-01194-8. PMID 35164805